CLINICAL TRIAL: NCT06858813
Title: A Phase 1 First-in-Human Study Evaluating Safety, Pharmacokinetics and Efficacy of ABBV 324 in Adults With Hepatocellular Cancer or Squamous Cell Non-Small Cell Lung Cancer
Brief Title: A Study to Assess Adverse Events and Change in Disease Activity of Intravenously (IV) Infused ABBV-324 in Adult Participants With Hepatocellular Cancer (HCC) or Squamous-Cell Non-Small Cell Lung Cancer (LUSC)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M25-292; 2024-518012-39 (Other: EU CT)
Record Dates: First submitted 2025-02-28; First posted 2025-03-05 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Hepatocellular Cancer; Squamous-Cell Non-Small Cell Lung Cancer
Keywords: Hepatocellular Cancer; Squamous-Cell Non-Small Cell Lung Cancer; LUSC; HCC; ABBV-324; Lenvatinib
MeSH Terms: conditions — Liver Neoplasms | interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Part 1 Dose Escalation: ABBV-324 (Experimental): Participants will receive escalating doses of ABBV-324 as part of the approximately 6.5 year study duration.
  Interventions: Drug: ABBV-324
- Part 2 Dose Optimization Arm 1: ABBV-324 Dose 1 (Experimental): Participants will receive ABBV-324 dose 1 as part of the approximately 6.5 year study duration.
  Interventions: Drug: ABBV-324
- Part 2 Dose Optimization Arm 1: ABBV-324 Dose 2 (Experimental): Participants will receive ABBV-324 dose 2 as part of the approximately 6.5 year study duration.
  Interventions: Drug: ABBV-324
- Part 2 Dose Optimization Arm 1: ABBV-324 Dose 3 (Experimental): Participants will receive ABBV-324 dose 3 as part of the approximately 6.5 year study duration.
  Interventions: Drug: ABBV-324
- Part 2 Comparator Arm 4: Lenvatinib (Active Comparator): Participants will receive lenvatinib as part of the approximately 6.5 year study duration.
  Interventions: Drug: Lenvatinib

INTERVENTIONS:
Drug: Lenvatinib — Oral Capsule
  Arms: Part 2 Comparator Arm 4: Lenvatinib
Drug: ABBV-324 — Intravenous (IV) Infusion
  Arms: Part 1 Dose Escalation: ABBV-324; Part 2 Dose Optimization Arm 1: ABBV-324 Dose 1; Part 2 Dose Optimization Arm 1: ABBV-324 Dose 2; Part 2 Dose Optimization Arm 1: ABBV-324 Dose 3

SUMMARY:
HCC is a common cancer worldwide and a leading cause of cancer-related death. Lung cancer is the most frequently diagnosed cancer in the world, and the leading cause of cancer deaths. The purpose of this study is to assess adverse events and change in disease activity when ABBV-324 is given to adult participants to treat hepatocellular cancer (HCC) or squamous-cell non-small cell lung cancer (LUSC).

ABBV-324 is an investigational drug being developed for the treatment of HCC and LUSC. Study doctors put the participants in groups called arms. Each arm receives ABBV-324 alone (monotherapy) or a comparator drug, lenvatinib followed by a safety follow-up period. Approximately 232 HCC or LUSC will be enrolled in the study in approximately 45 sites worldwide.

In the dose escalation stage participants will be treated with increasing intravenous (IV) doses of ABBV-324 until the dose reached is tolerable and expected to be efficacious. In the dose optimization stage participants will receive ABBV-324, or a comparator of oral lenvatinib. The study will run for a duration of approximately 6.5 years.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at an approved institution (hospital or clinic). The effect of the treatment will be frequently checked by medical assessments, blood tests, questionnaires and side effects.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Hepatocellular cancer (HCC) only: Child-Pugh A classification within 7 days before Cycle 1, Day 1 dosing.
* Laboratory values meeting the criteria outlined in the protocol.
* QT interval corrected for heart rate (QTc) < 470 msec (using Fridericia's correction), no Grade 3 arrythmia, and no other clinically significant cardiac abnormalities.
* Measurable disease per RECIST version 1.1.
* Part 1 and Part 2 - participants with HCC meeting the following disease activity criteria:

  * Locally advanced or metastatic and/or unresectable HCC with diagnosis confirmed by histology or cytology. Participants with fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma/HCC are not eligible to enroll.
  * Disease that is not amenable to surgical and/or locoregional therapies, or progressive disease after surgical and/or locoregional therapies. For participants who progressed after locoregional therapy for HCC, locoregional therapy must have been completed >= 28 days prior to baseline scan for the current study.
  * Part 1: Failure of at least 1 prior systemic treatment for HCC.
  * Part 2: Failure of at least 1 prior systemic treatment consisting of an immune checkpoint inhibitor (CPI) containing regimen for HCC, including but not limited to, atezolizumab in combination with bevacizumab or tremelimumab in combination with durvalumab. Note: Participants who have received prior lenvatinib will not be eligible for Part 2.
* Part 1 only - participants with squamous-cell non-small cell lung cancer (LUSC) meeting the following disease activity criteria:

  * Advanced or metastatic LUSC that is not amenable to surgical resection.
  * Must have failed at least 1 prior line of therapy that included at least platinum-based chemotherapy and an immune CPI, and/or an appropriate targeted therapy (if applicable), or is not suitable for other approved therapeutic options that have demonstrated clinical benefit at the judgment of the investigator. Participants should have no more than 2 lines of prior cytotoxic chemotherapy excluding neoadjuvant and/or adjuvant. Participants who are intolerant of standard therapy are eligible.

Exclusion Criteria:

* Unresolved clinically significant adverse events (AEs) > Grade 1 from prior anticancer therapy except for alopecia.
* Untreated brain or meningeal metastases (i.e., participants with history of metastases are eligible provided they do not require ongoing steroid treatment for cerebral edema and have shown clinical and radiographic stability for at least 14 days after definitive therapy). Participants may continue with antiepileptic therapy if required.
* History of interstitial lung disease (ILD) or pneumonitis that required treatment with systemic steroids, nor any evidence of active ILD or pneumonitis on screening chest computed tomography (CT) scan.
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis.
* History of clinically significant, intercurrent lung-specific illnesses including, but not limited to:

  * Underlying pulmonary disorder (i.e., pulmonary emboli within 3 months of the study enrollment, severe asthma, severe COPD, restrictive lung disease, pleural effusion, dependence on supplemental oxygen, etc.).
  * Any autoimmune, connective tissue or inflammatory disorders with documented or suspicious pulmonary involvement at Screening.
* Must have discontinued anticancer therapy with antineoplastic intent including chemotherapy, radiation therapy, immunotherapy, biologic, or any investigational therapy within 14 days or 5 half lives of the drug (whichever is shorter) prior to the first dose of ABBV-324. Palliative radiation therapy for bone, skin or subcutaneous metastases with 10 fractions or less is permitted and not participant to a washout period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2030-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AE)s | Up to Approximately 4 Years
  An adverse event is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Number of Participants with Change in Vital Signs | Up to Approximately 4 Years
  Number of Participants with Change in Vital Signs will be assessed.
Number of Participants with Change in Electrocardiogram (ECG) | Up to Approximately 4 Years
  Number of Participants with Change in ECG will be assessed.
Number of Participants with Change in Clinical Laboratory Tests | Up to Approximately 4 Years
  Number of participants with change in clinical laboratory tests will be assessed.
Objective Response Rate (ORR) | Up to Approximately 4 Years
  ORR is defined as the percentage of participants with a confirmed Complete Response or partial response(PR) per investigator review according to response evaluation criteria in solid tumors (RECIST) version 1.1.

SECONDARY OUTCOMES:
Area Under the Serum Concentration Versus Time Curve (AUC) of ABBV-324 | Up to Approximately 4 Years
  AUC of ABBV-324.
Maximum Observed Serum Concentration (Cmax) of ABBV-324 | Up to Approximately 4 Years
  Cmax of ABBV-324.
Time to Maximum Observed Serum Concentration (Tmax) of ABBV-324 | Up to Approximately 4 Years
  Tmax of ABBV-324.
Terminal Elimination Half-Life (t1/2) of ABBV-324 | Up to Approximately 4 Years
  t1/2 of ABBV-324.
Antidrug Antibody (ADA) | Up to Approximately 4 Years
  Incidence and concentration of anti-drug antibodies.
Neutralizing Antidrug Antibody (nADA) | Up to Approximately 4 Years
  Incidence and concentration of neutralizing anti-drug antibodies.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (21):
- United States (10):
  - City of Hope National Medical Center /ID# 270526, Duarte, California
  - City of Hope - Orange County Lennar Foundation Cancer Center /ID# 276120, Irvine, California
  - USC Norris Comprehensive Cancer Center /ID# 271573, Los Angeles, California
  - UC Irvine Medical Center /ID# 270507, Orange, California
  - UCLA - Santa Monica /ID# 275995, Santa Monica, California
  - University of Chicago Medical Center /ID# 270517, Chicago, Illinois
  - Washington University /ID# 275757, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center /ID# 271228, New York, New York
  - Thomas Jefferson University Sidney Kimmel Cancer Center /ID# 276269, Philadelphia, Pennsylvania
  - SCRI Oncology Partners /ID# 272750, Nashville, Tennessee
- China (2):
  - Nanfang Hospital - Southern Medical University /ID# 276916, Guangzhou, Guangdong
  - Zhongshan Hospital /ID# 276917, Shanghai, Shanghai Municipality
- Israel (3):
  - Rambam Health Care Campus /ID# 270604, Haifa
  - Hadassah Medical Center-Hebrew University /ID# 271235, Jerusalem
  - Rabin Medical Center /ID# 271236, Petah Tikva
- Japan (3):
  - National Cancer Center Hospital East /ID# 270585, Kashiwa-shi, Chiba
  - Kansai Medical University Hospital /ID# 272884, Hirakata-shi, Osaka
  - National Cancer Center Hospital /ID# 270583, Chuo-Ku, Tokyo
- Fdi Clinical Research /ID# 272960, San Juan, Puerto Rico
- Spain (2):
  - Hospital Universitario Fundación Jiménez Díaz /ID# 272718, Madrid
  - Hospital Universitario HM Sanchinarro /ID# 272719, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M25-292